CLINICAL TRIAL: NCT05573451
Title: CANNES (Cervical Cancer Lymph Node Staging): a Prospective, Imaging Study to Compare the Diagnostic Accuracy of Ultrasound, MRI and PET/CT in the Preoperative Assessment of Lymph Nodes in Cervical Cancer.
Brief Title: Comparison of the Accuracy of US, MRI and PET/CT in the Assessment of LNs in Cervical Cancer.
Acronym: CANNES
Status: Active, not recruiting | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Filip Fruhauf, Principial Investigator, General University Hospital, Prague
Other Study IDs: NU21-03-00461
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Lymph Node Metastasis; Cervical Cancer
MeSH Terms: conditions — Lymphatic Metastasis; Uterine Cervical Neoplasms | interventions — Positron Emission Tomography Computed Tomography; Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: ultrasound - transvaginal/transrectal + transabdominal — Each patient undergoes at least ultrasound examination and PET-CT.
  Other Names: PET-CT (positron emission tomography - computed tomography); DW-MRI (diffusion weighted magnetic resonance imaging)

SUMMARY:
Lymph node involvement is the most important negative prognostic factor in cervical cancer. Reliable preoperative lymph node assessment is of utmost importance to tailor the treatment. According to the current European guidelines local extent of the disease can be assessed by magnetic resonance imaging (MRI) or by ultrasound (US), if performed by properly trained sonographer. Positron emission tomography combined with computed tomography (PET/CT) is used as a reference standard for preoperative evaluation of lymph nodes. Another technique to assess nodes combining morphological and functional characteristics is diffusion-weighted MRI (DW/MRI). While US is considered the adequate alternative to MRI in local staging of cervical cancer, there is no relevant evidence of diagnostic performace of US in nodal assessment. However, retrospective analysis of diagnostic accuracy of US from our site brought promising results. Furthermore, there are no trials prospectively investigating these three imaging methods in the same study population. The CANNES study is a prospective multicenter trial comparing diagnostic accuracy of US, PET/CT and DW/MRI in preoperative assessment of pelvic lymph nodes in cervical cancer. The study is designed to establish new standard in preoperative assessment of pelvic lymph nodes in patients with cervical cancer. Ninety-one patients will be enrolled into the study within 36 months and each of them will undergo all three imaging methods. To avoid a bias all imaging examinations will be conducted independently and blinded among sonographers, radiologists and nuclear medicine physicians. By contrast, each surgeon will have all reports from imaging available before procedure to be used as a navigation. Surgical procedures will include sentinel lymph node biopsy, debulking/sampling or systematic dissection of pelvic nodes following current European guidelines.

DETAILED DESCRIPTION:
CANNES is a single arm, multicenter, prospective imaging trial. Patients referred with histopathologically confirmed cervical cancer will be clinically examined. As standard of care one of imaging method will be performed in preoperative local work-up - ultrasound or DW/MRI. The preference of imaging method of the first choice depends on the institutional practice. Eligible women meeting all inclusion criteria will be provided with the following documents ("Informed consent" and "Information for patients") and the objectives and the course of the study will be discussed with them. After the written consent, patients will be registered into the database using REDCap (Research Electronic Data Capture, www.project-redcap.org) electronic data capture tool. It is a secure, web-based application with controlled access designed to support data capture for research studies, hosted at MD Anderson.

To avoid any bias all imaging examinations will be conducted independently and blinded among sonographers, radologists and nuclear medicine physicians, i.e. without access to the reports from other examinations. In situation that sonographer is gynecologic oncologist, she/he will never perform and report ultrasound and surgery of the same patient. The same radiologist will never report the PET/CT and DW/MRI of the same patient. Examinators performing ultrasound scan and radiologists performing PET/CT or DW/MRI will be well instructed about standardized approach and evaluation of the imaging will follow predefined protocols. If a patient already had PET/CT or DW/MRI done by the referring hospital, the study radiologists decide about the quality of imaging and necessity to repeat them. All scans must be assessed by the radiologists involved in the study. Similarly, ultrasound examination will be only performed by expert sonographers participating in the trial. For every examination, a separate evaluation form (US form, PET/CT form and DW/MRI form) containing only the information of this examination will be used.

Surgery (laparoscopy, laparotomy or robotic surgery) should always be performed within 6 weeks after the first imaging method. Surgical procedure must include SLNB or sampling/debulking of suspicious/enlarged pelvic lymph nodes (± inframesenteric PALND) or systematic PLND. Surgeons will have all reports from ultrasound, PET/CT and DW/MRI available before surgery to be used as a navigation. All radiologically positive lymph nodes must be removed. Surgery evaluation form with precise description of the intraoperative finding will be filled in. Five evaluation forms will be completed (clinical data, US, PET/CT, DW/MRI, surgery) immediately when procedure finished using electronic database. The sixth evaluation form (pathology) will be completed when available by principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically verified cervical cancer
* FIGO stage IA1 L1 (lymphovascular space involvement) - IIIC2
* Patient eligible for surgery (PLND, sampling or debulking of LNs, SLNB)
* PET/CT scan not contraindicated
* 18 > Age < 80
* Eastern Cooperative Oncology Group (ECOG) performance status grade < 3
* Non-pregnant patient
* Informed consent signed

Exclusion Criteria:

* Tumor type other than primary cervical carcinomas
* Second malignant tumor under treatment
* FIGO stage IV (local spread to rectum or bladder, distant metastases)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histopathologically confirmed cervical cancer will be clinically examined. As standard of care one of imaging method will be performed in preoperative local work-up - ultrasound or DW/MRI. Per protocol PET/CT will be added.
  Surgery (laparoscopy, laparotomy or robotic surgery) should always be performed within 6 weeks after the first imaging method. Surgical procedure must include SLNB or sampling/debulking of suspicious/enlarged pelvic lymph nodes (± inframesenteric PALND) or systematic PLND. Surgeons will have all reports from ultrasound, PET/CT and DW/MRI available before surgery to be used as a navigation.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is comparison of the overall accuracy of ultrasound, PET/CT and DW/MRI in preoperative detection of pelvic lymph node macrometastases. | 36 months
  Sensitivity, specificity, PPV, NPV, overall acuracy, AUC, LR+, LR- and p-value will be calculated for each imaging method per patient and per site (separately right and left pelvic lymph nodes).

SECONDARY OUTCOMES:
Comparison of overall accuracy of US, PET/CT and DW/MRI in detection of pelvic lymph node involvement according to the TNM and FIGO classification (including both macrometastases and micrometastases) | 36 months
  Sensitivity, specificity, PPV, NPV, overall acuracy, AUC, LR+, LR- and p-value will be calculated for each imaging method per patient and per site (separately right and left pelvic lymph nodes).
Comparison of overall accuracy of US, PET/CT and DW/MRI in assessment of para-aortic lymph node involvement. | 36 months
  Sensitivity, specificity, PPV, NPV, overall acuracy, AUC, LR+, LR- and p-value will be calculated for each imaging method per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Fruhauf, Principal Investigator — General University Hospital
Locations (1):
- General University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No